CLINICAL TRIAL: NCT05890157
Title: Treatment Of Shallow Periodontal Pockets Using PRF As an Adjunct To Scaling And Root Planing In Periodontitis Patients, Randomized Clinical Trial
Brief Title: Treatment Of Shallow Periodontal Pockets Using PRF As an Adjunct To Scaling And Root Planing In Periodontitis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Sarah Alrihaymee, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRF as adjunct to ScRp
Record Dates: First submitted 2023-05-16; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test ScRp+PRF (Experimental): This site will treated by ScRp+PRF
  Interventions: Other: PRF
- Control ScRp (No Intervention): This site will treated by ScRp only

INTERVENTIONS:
Other: PRF — Split mouth randomized clinical trial will be the design of the study. 12 periodontitis patients with 24 opposite shallow periodontal pockets (4-6 mm in depth) will be selected. Randomization in this study will be achieved using toss of coin method in which periodontal pockets were designated either control site or test site. PRF will be used as an adjunct to scaling and root planing to treat the test sites. While control sites will be treated by scaling and root planing only. Clinal periodontal parameters will be recorded and GCF level of PDGF-BB will be measured at baseline and1- and 3- month follow-up visits to evaluate the healing response to the treatment.
  Arms: Test ScRp+PRF

SUMMARY:
Platelet rich fibrin (PRF) has been widely used in regenerative dentistry since it provides plenty amount of growth factors that enhance wound healing and tissue regeneration. Platelet derived growth factor-BB (PDGF-BB) is a growth factor with essential functions such as regulation of cell migration, proliferation, and differentiation. This study aims to evaluate the efficacy of PRF in improving the clinical periodontal parameters and GCF level of PDGF-BB.

DETAILED DESCRIPTION:
Split mouth randomized clinical trial is the design of the study. 12 periodontitis patients with 24 opposite shallow periodontal pockets (4-6 mm in depth) will be selected. Randomization in this study will be achieved using toss of coin method in which periodontal pockets will be designated either control site or test site. PRF will be used as an adjunct to scaling and root planing to treat the test sites. While control sites were treated by scaling and root planing only. Clinal periodontal parameters were recorded and GCF level of PDGF-BB will be measured at baseline and1- and 3- month follow-up visits to evaluate the healing response to the treatment.

ELIGIBILITY:
Inclusion Criteria:

•periodontitis

Exclusion Criteria:

* Periodontal therapy for the last 3 months
* Medical history of systemic diseases such as diabetes.
* Patients wearing dental prosthesis
* Alcoholic patients
* Teeth with grade II mobility, endodontic lesions, and teeth with untreated caries

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical attachment level | Change from baseline to 1-month and change from baseline to 3-month
  Using UNC-15 periodontal probe measured in mm
Change in Periodontal pocket depth measured in mm | Change from baseline to 1-month and change from baseline to 3-month
  Using UNC-15 periodontal probe measured in mm

SECONDARY OUTCOMES:
Change in plaque index | Change from baseline to 1-month and change from baseline to 3-month
  Using Sinless and Loe 1964 plaque index scores
Change in bleeding on probing percentage | Change from baseline to 1-month and change from baseline to 3-month
  Using UNC-15 periodontal probe
Change in GCF level of platelet derived growth factor | Change from baseline to 1-month and change from baseline to 3-month
  Using periocol paper to collect GCF and analysed by ELISA test

IPD SHARING:
Plan to Share IPD: Undecided